CLINICAL TRIAL: NCT07359755
Title: A Comparative Analysis of Vaginal Mesh Surgery Versus Robotic-assisted Abdominal Mesh Surgery in the Treatment of Apical Genital Prolapse: a Prospective Randomized Non-inferiority Study.
Brief Title: Vaginal Mesh Surgery Versus Robotic-assisted Abdominal Mesh Surgery in the Treatment of Apical Prolapse - Prospective Randomized Non-inferiority Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcelo Hisano, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7.815.545; 86242424.1.0000.0068 (Registry Identifier: CAAE)
Record Dates: First submitted 2025-11-30; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Pelvic Organ Prolapse (POP); Pelvic Organ Prolapse Vaginal Surgery; Mesh Reinforcement; Vaginal Apex/Uterine Prolapse
Keywords: Pelvic organ prolapse; Vaginal prolapse; Vaginal mesh; Robotic-assisted sacrocolpopexy; Sacrocolpopexy; Uterine prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse; Uterine Prolapse

STUDY DESIGN:
Intervention Model Description: This prospective, randomized trial is designed to evaluate the treatment of apical vaginal prolapse, with the objective of demonstrating the non-inferiority of vaginal mesh repair compared to robotic-assisted abdominal sacral colpopexy. The assessment will focus on objective cure rates as well as secondary outcomes, including clinical complications, mesh erosion, and patient-reported clinical improvements measured through validated questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vaginal mesh surgery (Experimental): Vaginal mesh surgery for apical prolapse
  Interventions: Procedure: Vaginal mesh surgery for apical prolapse
- Robotic-assited abdominal sacrocolpopexy (Active Comparator): Robotic-assisted abdominal mesh surgery with Upsylon device (Boston Scientific - USA) for vaginal apical prolapse
  Interventions: Procedure: Robotic-assisted abdominal mesh surgery with Upsylon device (Boston Scientific - USA) for vaginal apical prolapse

INTERVENTIONS:
Procedure: Vaginal mesh surgery for apical prolapse — Cirurgia com tela vaginal para prolapso apical.
  Arms: Vaginal mesh surgery
Procedure: Robotic-assisted abdominal mesh surgery with Upsylon device (Boston Scientific - USA) for vaginal apical prolapse — Cirurgia robótica assistida por tela abdominal com dispositivo Upsylon (Boston Scientific - EUA) para prolapso apical vaginal.
  Arms: Robotic-assited abdominal sacrocolpopexy

SUMMARY:
The goal of this study is to compare vaginal mesh surgery with abdominal robotic-assisted mesh surgery for the treatment of genital prolapse in women. The main questions it seeks to answer are:

* Is the objective cure rate for vaginal mesh surgery non-inferior to that of the abdominal approach?
* Is the use of vaginal mesh as safe as abdominal mesh?

DETAILED DESCRIPTION:
This is a prospective, randomized non-inferiority study designed to compare the objective outcomes of treating apical compartment pelvic organ prolapse (POP) using robot-assisted abdominal mesh surgery versus vaginal mesh surgery. Additionally, clinical parameters such as mesh erosion, pain, and symptom-specific quality of life will be assessed utilizing an internationally validated instrument adapted for Portuguese-speaking populations.

Patients diagnosed with stage II or higher apical compartment pelvic organ prolapse (POP), with or without a uterus, who require surgical intervention and provide informed consent will be randomized through REDCap® software to determine the surgical approach.

The interventions under investigation include: vaginal prolapse repair with placement of the Splentis® mesh (Promedon®, Córdoba, Argentina) - not FDA approved, comprising anterior colporrhaphy combined with suspension of the cervix or vaginal vault, with bilateral anchoring of the mesh to the sacrospinous ligaments; and robot-assisted laparoscopic abdominal repair employing the Upsylon® mesh (Boston Scientific®, USA) - FDA approved - via colpocervicopexy, involving mesh fixation to the anterior and superior vaginal walls as well as the sacral promontory.

The sample size was calculated to assess the non-inferiority of the vaginal approach compared with the abdominal approach. Assuming an objective cure rate (stage 0 or I) of 90% for the abdominal group and 80% for the vaginal group, with a two-sided significance level of p < 0.05 and an anticipated loss to follow-up of up to 10% in each group, a minimum of 43 participants per arm (total of 86 patients) was required. The calculation was based on detecting a non-inferiority margin considered clinically acceptable for the primary outcome.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients diagnosed with apical compartment genital prolapse of stage II or higher, who have an indication for surgical correction.

Exclusion Criteria:

* The following exclusion criteria will apply: patients who are unable or unwilling to complete validated outcome assessment instruments; those requiring concomitant surgical procedures (e.g., hysterectomy or any other intervention that may alter pelvic floor anatomy);
* individuals with a prior history of pelvic radiotherapy;
* patients with congenital or acquired anomalies of the urogenital or gastrointestinal systems;
* and those with medical conditions that constitute a contraindication to elective surgical intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Objective Cure Rate | Patients will undergo evaluations at 1 month postoperatively and subsequently at 6-month intervals from the date of surgery, continuing until 24 months of follow-up have been completed.
  The criteria for objective cure will be defined according to the Pelvic Organ Prolapse Quantification (POP-Q) system, with point C positioned at -6 cm or higher (proximal), corresponding to stage 0 or I genital prolapse.

SECONDARY OUTCOMES:
Surgical complication | Patients will undergo evaluations at 1 month postoperatively and subsequently at 6-month intervals from the date of surgery, continuing until 24 months of follow-up have been completed.
  Complications will be evaluated in the perioperative period and during follow-up, encompassing surgical complications, long-term adverse events such as mesh erosion, and complications necessitating corrective interventions. These complications will be categorized according to the Clavien-Dindo classification system.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clinicas da Faculdade de Medicina de Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol; Statistical Analysis Plan (SAP)
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bataller E, Ros C, Angles S, Gallego M, Espuna-Pons M, Carmona F. Anatomical outcomes 1 year after pelvic organ prolapse surgery in patients with and without a uterus at a high risk of recurrence: a randomised controlled trial comparing laparoscopic sacrocolpopexy/cervicopexy and anterior vaginal mesh. Int Urogynecol J. 2019 Apr;30(4):545-555. doi: 10.1007/s00192-018-3702-7. Epub 2018 Jul 9. PMID 29987345
- [Background] Lee RK, Mottrie A, Payne CK, Waltregny D. A review of the current status of laparoscopic and robot-assisted sacrocolpopexy for pelvic organ prolapse. Eur Urol. 2014 Jun;65(6):1128-37. doi: 10.1016/j.eururo.2013.12.064. Epub 2014 Jan 8. PMID 24433811
- [Background] Coolen AWM, Bui BN, Dietz V, Wang R, van Montfoort APA, Mol BWJ, Roovers JWR, Bongers MY. The treatment of post-hysterectomy vaginal vault prolapse: a systematic review and meta-analysis. Int Urogynecol J. 2017 Dec;28(12):1767-1783. doi: 10.1007/s00192-017-3493-2. Epub 2017 Oct 16. PMID 29038834
- [Background] Maher CF, Feiner B, DeCuyper EM, Nichlos CJ, Hickey KV, O'Rourke P. Laparoscopic sacral colpopexy versus total vaginal mesh for vaginal vault prolapse: a randomized trial. Am J Obstet Gynecol. 2011 Apr;204(4):360.e1-7. doi: 10.1016/j.ajog.2010.11.016. PMID 21306698
- [Background] Hudson CO, Northington GM, Lyles RH, Karp DR. Outcomes of robotic sacrocolpopexy: a systematic review and meta-analysis. Female Pelvic Med Reconstr Surg. 2014 Sep-Oct;20(5):252-60. doi: 10.1097/SPV.0000000000000070. PMID 25181374
- [Background] Rovner E, Chermansky C, Costantini E, Dmochowski R, Enemchukwu E, Ginsberg DA, Heesakkers J, Menefee S, Nadeau G, Rardin C, Zimmern P. Recommendations of the SUFU/AUGS/ICS Female Stress Urinary Incontinence Surgical Publication Working Group: A common standard minimum data set for the literature. Neurourol Urodyn. 2024 Nov;43(8):1753-1764. doi: 10.1002/nau.25445. Epub 2024 Jun 5. PMID 38837735
- [Background] Peterson TV, Pinto RA, Davila GW, Nahas SC, Baracat EC, Haddad JM. Validation of the Brazilian Portuguese version of the pelvic floor bother questionnaire. Int Urogynecol J. 2019 Jan;30(1):81-88. doi: 10.1007/s00192-018-3627-1. Epub 2018 Mar 16. PMID 29549393
- [Background] Angelo PH, de Queiroz NA, Leitao ACR, Marini G, Micussi MT. Validation of the international consultation on incontinence modular questionnaire - female lower urinary tract symptoms (ICIQ-FLUTS) into brazilian portuguese. Int Braz J Urol. 2020 Jan-Feb;46(1):53-59. doi: 10.1590/S1677-5538.IBJU.2019.0234. PMID 31851458
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Kisby CK, Occhino JA, Bews KA, Habermann EB, Linder BJ. Perioperative Complications in Minimally Invasive Sacrocolpopexy Versus Transvaginal Mesh in the Management of Pelvic Organ Prolapse: Analysis of a National Multi-institutional Dataset. Female Pelvic Med Reconstr Surg. 2021 Feb 1;27(2):72-77. doi: 10.1097/SPV.0000000000000738. PMID 31094716
- [Background] Maher CF, Baessler KK, Barber MD, Cheong C, Consten ECJ, Cooper KG, Deffieux X, Dietz V, Gutman RE, van Iersel JJ, Nager CW, Sung VW, de Tayrac R. Surgical management of pelvic organ prolapse. Climacteric. 2019 Jun;22(3):229-235. doi: 10.1080/13697137.2018.1551348. Epub 2018 Dec 21. PMID 30572743
- [Background] Haylen BT, Maher CF, Barber MD, Camargo S, Dandolu V, Digesu A, Goldman HB, Huser M, Milani AL, Moran PA, Schaer GN, Withagen MI. An International Urogynecological Association (IUGA) / International Continence Society (ICS) Joint Report on the Terminology for Female Pelvic Organ Prolapse (POP). Neurourol Urodyn. 2016 Feb;35(2):137-68. doi: 10.1002/nau.22922. Epub 2016 Jan 7. PMID 26749391
- [Background] Maher C, Yeung E, Haya N, Christmann-Schmid C, Mowat A, Chen Z, Baessler K. Surgery for women with apical vaginal prolapse. Cochrane Database Syst Rev. 2023 Jul 26;7(7):CD012376. doi: 10.1002/14651858.CD012376.pub2. PMID 37493538
- [Background] Zhang CY, Sun ZJ, Yang J, Xu T, Zhu L, Lang JH. Sacrocolpopexy compared with transvaginal mesh surgery: a systematic review and meta-analysis. BJOG. 2021 Jan;128(1):14-23. doi: 10.1111/1471-0528.16324. Epub 2020 Jun 15. PMID 32426903
- [Background] Nygaard I, Bradley C, Brandt D; Women's Health Initiative. Pelvic organ prolapse in older women: prevalence and risk factors. Obstet Gynecol. 2004 Sep;104(3):489-97. doi: 10.1097/01.AOG.0000136100.10818.d8. PMID 15339758
- [Background] Hendrix SL, Clark A, Nygaard I, Aragaki A, Barnabei V, McTiernan A. Pelvic organ prolapse in the Women's Health Initiative: gravity and gravidity. Am J Obstet Gynecol. 2002 Jun;186(6):1160-6. doi: 10.1067/mob.2002.123819. PMID 12066091
- [Background] Handa VL, Garrett E, Hendrix S, Gold E, Robbins J. Progression and remission of pelvic organ prolapse: a longitudinal study of menopausal women. Am J Obstet Gynecol. 2004 Jan;190(1):27-32. doi: 10.1016/j.ajog.2003.07.017. PMID 14749630
- [Background] Bradley CS, Zimmerman MB, Qi Y, Nygaard IE. Natural history of pelvic organ prolapse in postmenopausal women. Obstet Gynecol. 2007 Apr;109(4):848-54. doi: 10.1097/01.AOG.0000255977.91296.5d. PMID 17400845

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-09-03): https://cdn.clinicaltrials.gov/large-docs/55/NCT07359755/SAP_000.pdf